CLINICAL TRIAL: NCT05387863
Title: Evaluation of a Decision Aid in the Treatment Planning of Small Renal Tumors
Brief Title: Decision Aid (DA) for Renal Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-01670
Record Dates: First submitted 2022-05-19; First posted 2022-05-24 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Kidney Tumor; Renal Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decision Aid (DA) Web Tool (Experimental)
  Interventions: Other: Decision Aid (DA) Web Tool
- Institutional Pamphlet (Active Comparator)
  Interventions: Other: Institutional Pamphlet

INTERVENTIONS:
Other: Decision Aid (DA) Web Tool — The DA web tool provides information on kidney masses and available treatment options. It uses risk communication, directed teaching, and interactive benefit-harm assessment to present information.
  Arms: Decision Aid (DA) Web Tool
Other: Institutional Pamphlet — The institutional pamphlet provides information on kidney masses, but does not use risk communication, directed teaching, or interactive benefit-harm assessment.
  Arms: Institutional Pamphlet

SUMMARY:
The objective of this study is to understand how patients make decisions about treating their kidney masses, and to identify key values and preferences for treating their kidney masses. The study team will develop a decision aid (DA) using the decision-analytic model to communicate personalized benefit/harm estimates to patients and promote patient-centered treatment of renal tumors.

ELIGIBILITY:
Inclusion Criteria:

* Male and female post-op and pre-op patients, ages 18 and older, diagnosed with a localized renal tumor up to 4 cm in diameter.
* Patients scheduled for standard-of-care clinical exams with the NYU Urology Department

Exclusion Criteria:

* Stage IV cancer of any type
* Inability to provide informed consent
* Vulnerable subjects will not be recruited

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Knowledge Score | Pre-Counsel, 1 day Visit
  Via a survey, patients will be asked general questions about kidney masses and their treatments. There are 10 questions, each scored as correct or incorrect (0 or 1), and the last question has 3 sub-components each scored 0-1. The total range of score is 0-10; a score of 10 indicates strongest knowledge on kidney masses/treatments.
Decision Satisfaction Score | Post-Counsel, 1 day Visit
  Via a survey, patients provide their opinion on 16 statements. Each statement is scored 1 (strongly disagree) to 5 (strongly agree). The total range of score is 1-80; a higher score indicates higher satisfaction.
Shared Decision Making | Post-Counsel, 1 day Visit
  This is a binary outcome measure. Patients will be asked whether or not they felt they participated in a shared decision making process: 0 for no, 1 for yes.

CONTACTS AND LOCATIONS:
Overall Officials: Stella Kang, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data upon reasonable request. Requests should be directed to stella.kang@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Fogarty J, Siriruchatanon M, Makarov D, Langford A, Kang S. An Evaluation of a Web-Based Decision Aid for Treatment Planning of Small Kidney Tumors: Pilot Randomized Controlled Trial. JMIR Res Protoc. 2022 Sep 2;11(9):e41451. doi: 10.2196/41451. PMID 36053558